CLINICAL TRIAL: NCT03912181
Title: Medical Complications in Familial and Multifactorial Chylomicronaemia Syndromes From a 10 Year Follow-up Linking Datasets Between Patient Medical Records and Patient Claims: the ESTHYM Study
Brief Title: Medical Complications in Familial and Multifactorial Chylomicronaemia Syndromes
Acronym: ESTHYM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0864
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Familial Chylomicronemia Syndrome; Multifactorial Chylomicronemia Syndrome
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Familial chylomicronaemia syndrome (FCS): * Patient homozygous or compound heterozygous mutation in lipoprotein lipase (LPL) gene
  * Patient homozygous or compound heterozygous mutation in any Apolipoprotein A5 (Apo A5), glycosylphosphatidylinositol anchored high density lipoprotein binding protein 1 (GPI HBP1), lipase maturation factor 1 (LMF1), Apolipoprotein C2 (ApoC2), genes and heterozygous (het) mutation in LPL gene
- Multifactorial chylomicronemia syndrome: * Patient with heterozygous mutation in lipoprotein lipase (LPL) , Apolipoprotein A5 (Apo AV), GPI HBP1, LMF1, ApoC2 genes and any additional combination of functional variant
  * Patient with any additional combination of functional variant in LPL gene Apo AV, glycosylphosphatidylinositol anchored high density lipoprotein binding protein 1 (GPI HBP1), lipase maturation factor 1 (LMF1), Apolipoprotein C2 (ApoC2) genes

SUMMARY:
A retrospective, systematic study of reimbursed healthcare costs over a 10 year period in patients suffering from Familial Chylomicronaemia Syndromes (FCS) or Multifactorial Chylomicronaemia Syndromes (MCS) in order to establish the relative healthcare burden of both syndromes by linking the Hospices Civils de Lyon (HCL) registry of FCS or MCS patients and data obtained from FCS or MCS patients followed in Paris, Nantes and Lyon to the French National Health System (NHS) healthcare claims database, the Système National d'Information Inter-Régimes de l'Assurance Maladie (SNIIR-AM).

A probabilistic approach will be used to link databases. This linkage will be based on the following variables: age, gender, date of discharge of any hospitalization, date of any imaging procedure.

This study will help to describe, in real life, the management of severe hyperglyceridaemia in France. In addition, the descriptive results will help obtain a better understanding of the patients suffering from this disease, the burden of the disease and the healthcare consumption linked to this disease. Even if this consumption of care has been relatively unexplored until this point, it is not negligible. The potential of merging genomics and claims data for cardiovascular research could help to identify ways to optimize disease

ELIGIBILITY:
Inclusion Criteria:

* genetically documented FCS
* genetically documented MCS

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients male or female at least 18 years old having genetically documented familial or multifactorial chylomicronaemia syndrome.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Acute Pancreatitis, Ischemic Cardiovascular Disease and any additional co-morbidity | 2006-2016 (10 year follow-up)
  outcomes obtained by anonymous linkage with the Système National des Données de Santé (SNDS) national data base of any health resource consumption (> 40x106 subjects exhaustive compilation, linkage with Programme de médicalisation des systèmes d'information (PMSI) (diagnosis data base) and death registry)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Moulin, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Derived] Belhassen M, Van Ganse E, Nolin M, Berard M, Bada H, Bruckert E, Krempf M, Rebours V, Valero R, Moulin P. 10-Year Comparative Follow-up of Familial versus Multifactorial Chylomicronemia Syndromes. J Clin Endocrinol Metab. 2021 Mar 8;106(3):e1332-e1342. doi: 10.1210/clinem/dgaa838. PMID 33221907